CLINICAL TRIAL: NCT05843084
Title: The STEREO-DBS Study: 7-Tesla MRI Brain Network Analysis for Deep Brain Stimulation
Acronym: STEREO-DBS
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Maarten Bot, Principal Investigator, Associative Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W20_540 # 20.599
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Diffusion Magnetic Resonance Imaging; Brain; Subthalamic Nucleus; Deep Brain Stimulation; Human; Treatment Outcome
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: 7T MRI network analysis for deep brain stimulation in Parkinson's disease — We hypothesize that the implementation of 7T MRI network analysis can enhance the effectiveness of DBS by improving motor symptoms and quality of life in PD patients.

SUMMARY:
Rationale: Deep brain stimulation (DBS) of the nucleus subthalamicus (STN) is an effective surgical treatment for the patients with advanced Parkinson's disease, despite optimal pharmacological treatment. However, individual improvement after DBS remains variable and 50% of patients show insufficient benefit. To date, DBS-electrode placement and settings in the highly connected STN are based on 1,5-Tesla or 3-Tesla MR-images. These low resolution and solely structural modalities are unable to visualize the multiple brain networks to this small nucleus and prevent electrode activation directed at its cortical projections. By using structural 7-Tesla MRI (7T MRI) connectivity to visualize (malfunctioning) brain networks, DBS-electrode placement and activation can be individualized.

Objective: Primary objective of the study is to determine whether visualisation of cortical projections originating in the STN and the position of the DBS electrode relative to these projections using 7T MRI improves motor symptoms as measured by the disease-specific Unified Parkinson's Disease Rating Scale (UPDRS-III).

Secondary outcomes are: disease related daily functioning, adverse effects, operation time, quality of life, patient satisfaction with treatment outcome and patient evaluation of treatment burden.

Study design: The study will be a single center prospective observational study.

Study population: Enrollment will be ongoing from April 2022. Intervention (if applicable): No intervention will be applied. Application of 7T MRI for DBS is standard care and outcome scores used will be readily accessible from the already existing advanced electronic DBS database.

Main study parameters/endpoints: The primary outcome measure is the change in motor symptoms as measured by the disease-specific Unified Parkinson's Disease Rating Scale (UPDRS-III). This is measured after 6 months of DBS as part of standard care. The secondary outcome measures are the Amsterdam Linear Disability Score for functional health status, Parkinson's Disease Questionnaire 39, Starkstein apathy scale, patient satisfaction with the treatment, patient evaluation of treatment burden, operating time, hospitalization time, change of tremor medication, side effects and complications.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The proposed observational research project involves treatment options that are standard care in daily practice. The therapies will not be combined with other research products. Participation in this study constitutes negligible risk according to NFU criteria for human research.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Deep brain stimulation for Parkinson's disease Deep brain stimulation (DBS) is an effective treatment in Parkinson's disease (PD), a debilitating neurological disorder. The effect of DBS relies on the modulation of malfunctioning brain networks by delivering electrical pulses within the subthalamic nucleus, deeply seated in the brainstem and the size of a few millimeters (STN; comparable to the size of a coffee bean). However, individual improvement after DBS remains variable and 50% of patients show insufficient benefit. By using structural 7-Tesla magnetic resonance imaging (7T MRI) connectivity to visualize malfunctioning networks, DBS-electrode placement and activation can be individualized.

Current DBS-electrode placement and settings in the highly connected STN are based on 1.5-Tesla or 3-Tesla MR-images. These low resolution modalities are unable to visualize the multiple brain networks to this small nucleus and prevent electrode activation directed at its cortical projections. Integrated structural (7T MRI) network maps will enable brain network-based and patient-specific DBS, improving motor symptoms and quality of life.

7T MRI brain network analysis Since the 1980s, DBS for PD was targeting the STN, a deep-seated grey matter brain nucleus. Current emphasis in the field of DBS is on neural networks rather than separate nuclei in the brain. Several studies showed PD to arise from pathological network activity in subthalamic-cortical projections. In recent years several DBS groups reported about using MRI connectivity to visualize the subthalamic-cortical projections, in DBS for PD.

The small STN is part of multiple large brain networks. DBS is effective in improving UDPRS and quality of life for PD patients only by modulating its motor network. For improving DBS placement and activation, it is essential to understand the networks and the modulatory effect of stimulation. Thus far, visualization of these networks was limited due to low resolution and the lack of structural connectivity (visualising subthalamic-cortical projections using diffusion weighted MRI and probabilistic connectivity).

The investigators therefore added 7T T2 and diffusion-weighted sequences at the Spinoza Centre and showed that probabilistic subthalamic network analyses (STN segmentation) successfully identifies the area within the STN that has the highest density of connections with the motor network in PD patients. In a recent pilot study the investigators showed the implementation of 7T MRI for STN segmentation is well suited within the existing surgical workflow. By generating a 7-Tesla MRI showing the STN (coloured) motor subdivision, this technique clearly visualized this new DBS target. The retrospective analysis showed for conventional MRI targeting strategies only a minority of DBS electrodes were placed in the motor STN. Moreover, the DBS electrodes that were placed in the motor STN resulted in a significantly higher mean improvement (80% versus 50%, measured by the UPDRS-III score).

Generating the 7T MRI network maps for DBS The STN and its cortical connections will be visualized using 7T T2-weighted and diffusion weighted imaging. Three major projections of the STN will be visualised: projections connecting to primary and supplementary motor cortex (motor), projections to the prefrontal cortex (associative) and projections to the basofrontal cortex (limbic). The location of the electrode (using computed tomography) will be visualised relative to the three segmented subdivisions of the STN.

The 7T MRI network map, generated by combining T2 and diffusion weighted MRI, shows the STN (coloured) subdivisions and their cortical projections. The result will then show in which STN subdivision(s) the DBS-electrode contact is situated and to which cortical area the STN subdivision projects. Clinical test scores of the electrode contact will then be correlated to the network maps. Stimulation parameters based on 7T MRI network maps are used to optimize and predict outcome in terms of beneficial clinical effects (suppression tremor, bradykinesia, rigidity) and side effects (speech, gait, apathy). As all network maps are visualised on MRI, this will readily enable both individual and group analyses (co-registrating maps of multiple patients).

Adverse effects In the 350 7T MR-scans the investigators have performed to date, we rarely encountered non-compatible implants or severe claustrophobia. Every patient undergoes screening with a MRI safety questionnaire and MRI metal detector (preventing taking ferromagnetic materials into the MRI). 7T MRI is a non-invasive technique which causes no pain and, importantly, the electromagnetic fields produce no known tissue damage of any kind. The MR system may make loud tapping, knocking, or other noises at times during the procedure. Earplugs are provided to prevent problems that may be associated with noise generated by the scanner. At all times, the patient will be (visually) monitored and will be able to communicate with the 7T MRI technologist using an intercom system. The patient may (request to) stop the acquisition at any time by using the push button (hold by the patient continuously).

In sum, due to implementation of 7T MRI brain network analysis, it is now possibly to directly visualize the motor part of the STN. In current observational study this technique will be evaluated in a prospective fashion, introducing patient specific brain network-guided DBS for PD with delivering a unique and hitherto unavailable dataset: 7T MRI visualizes the anatomical connections of the STN for each individual DBS electrode contact. Instead of a one-DBS-fits all model, the tailored network analyses enable personalized precision modelling in DBS.

ELIGIBILITY:
1.2 Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age > 18 years;
* Idiopathic PD who underwent STN DBS

1.3 Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Legally incompetent adults;
* No written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STUDY POPULATION 1.1 Population (base) Patients with advanced Parkinson's disease who underwent DBS electrode placement using 7T MRI network analysis. If the patient is eligible, the physician coordinating the study will inform the patient, hand over written information about the observational study, and subsequently ask the patient to consider participation. If the patient wants to participate, the informed consent form will be signed. Patients will be given as much time as needed to decide whether to participate in the study. Enrollment will be ongoing from April 2023; patients who underwent 7T MRI network analysis based DBS before this date will also be eligible to participate (all DBS patients are registered in the prospective electronic Castor database).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2033-04-11 (Estimated); Study Completion 2033-04-11 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS-III) | April 2022 - April 2033
  The amount of decrease in motor symptoms indicated by change in the disease-specific Unified Parkinson's Disease Rating Scale (UPDRS-III) after six months of deep brain stimulation. The UPDRS-III scores are between 7 and 86; higher scores indicating worse (more severe) motor symptoms.

SECONDARY OUTCOMES:
The Amsterdam Linear Disability Score for functional health status | April 2022 - April 2033
  The Amsterdam Linear Disability Score (ALDS) is a generic itembank which measures disability, as expressed by the ability to perform activities of daily living. These scores are linearly transformed into values between 0 and 100. Lower scores indicate more disability.
Parkinson's disease questionnaire-39 | April 2022 - April 2033
  The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. It also assesses the impact of Parkinson's on specific dimensions of functioning and wellbeing. The scores are between 0 and 100 (the sum of all 39 items), higher score indicating more health problems.
Starkstein apathy scale | April 2022 - April 2033
  The 14-item Starkstein Apathy Scale (SAS) is used to measure the severity of apathetic symptoms in Parkinson disease. The scores are between 0 and 42. Higher scores indicating worse apathy.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Bot, MD PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From april 2022

REFERENCES:
- [Background] 1. Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. Apr 9 2021. 2. Bot M, Schuurman PR, Odekerken VJJ, et al. Deep brain stimulation for Parkinson's disease: defining the optimal location within the subthalamic nucleus. J Neurol Neurosurg Psychiatry. May 2018;89(5):493-498. 3. Mathiopoulou V, Rijks N, Caan MWA, et al. Utilizing 7-Tesla Subthalamic Nucleus Connectivity in Deep Brain Stimulation for Parkinson Disease. Neuromodulation. Feb 22 2022. 4. Schrock LE, Patriat R, Goftari M, et al. 7T MRI and Computational Modeling Supports a Critical Role of Lead Location in Determining Outcomes for Deep Brain Stimulation: A Case Report. Front Hum Neurosci. 2021;15:631778. 5. Plantinga BR, Temel Y, Duchin Y, et al. Individualized parcellation of the subthalamic nucleus in patients with Parkinson's disease with 7T MRI. NeuroImage. Mar 2018;168:403-411. 6. Nowacki A, Barlatey S, Al-Fatly B, et al. Probabilistic Mapping Reveals Optimal Stimulation Site in Essential Tremor. Ann Neurol. May 2022;91(5):602-612. 7. Akram H, Sotiropoulos SN, Jbabdi S, et al. Subthalamic deep brain stimulation sweet spots and hyperdirect cortical connectivity in Parkinson's disease. NeuroImage. Sep 2017;158:332-345. 8. Jaradat A, Nowacki A, Montalbetti M, et al. Probabilistic Subthalamic Nucleus Stimulation Sweet Spot Integration Into a Commercial Deep Brain Stimulation Programming Software Can Predict Effective Stimulation Parameters. Neuromodulation. Feb 2023;26(2):348-355. 9. Rijks N, Potters WV, Dilai J, et al. Combining 7T T2 and 3T FGATIR: from physiological to anatomical identification of the subthalamic nucleus borders. J Neurol Neurosurg Psychiatry. Feb 19 2022. 10. Bot M, Verhagen O, Caan M, et al. Defining the Dorsal STN Border Using 7.0-T MRI: A Comparison to Microelectrode Recordings and Lower Field Strength MRI. Stereotact Funct Neurosurg. 2019;97(3):153-159.